CLINICAL TRIAL: NCT00004341
Title: Study of Genetic and Molecular Defects in Primary Immunodeficiency Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Washington (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11900; UW-533
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: X-Linked Agammaglobulinemia; X-Linked Hyper IgM Syndrome; Wiskott-Aldrich Syndrome; Leukocyte Adhesion Deficiency Syndrome
Keywords: Wiskott-Aldrich syndrome; X-linked agammaglobulinemia; X-linked hyper IgM syndrome; genetic diseases and dysmorphic syndromes; immunologic disorders and infectious disorders; leukocyte adhesion deficiency syndrome; primary immunodeficiency disease; rare disease
MeSH Terms: conditions — Bruton type agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome, Type 1; Wiskott-Aldrich Syndrome; Leukocyte-Adhesion Deficiency Syndrome; Genetic Diseases, Inborn; Immune System Diseases; Communicable Diseases; Primary Immunodeficiency Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Identify the molecular defects responsible for primary immunodeficiency disorders.

II. Explore the mutations within each syndrome to better understand the genetics of these disorders.

III. Study the function of the Wiskott-Aldrich syndrome proteins (WASP). IV. Design methods to identify carriers and for prenatal diagnosis. V. Explore new avenues for therapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are studied systematically to determine the extent of their immune deficiency and to confirm a specific diagnosis. Patients with a known immunodeficiency syndrome are studied in detail to identify the gene mutation, to assess the effect of the mutation on the gene product, and to establish cell lines for further in vitro assessment of the genetic defect. The function of Wiskott-Aldrich syndrome proteins (WASP) in hematopoietic cells is studied.

Family members of patients with X-linked disorders are studied to identify carrier females.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Primary immunodeficiency disease, e.g.: Leukocyte adhesion deficiency syndrome Wiskott-Aldrich syndrome X-linked agammaglobulinemia X-linked hyper IgM syndrome

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: Hans D. Ochs, Study Chair — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States

REFERENCES:
- [Background] Miki H, Nonoyama S, Zhu Q, Aruffo A, Ochs HD, Takenawa T. Tyrosine kinase signaling regulates Wiskott-Aldrich syndrome protein function, which is essential for megakaryocyte differentiation. Cell Growth Differ. 1997 Feb;8(2):195-202. PMID 9040941
- [Background] Zhu Q, Watanabe C, Liu T, Hollenbaugh D, Blaese RM, Kanner SB, Aruffo A, Ochs HD. Wiskott-Aldrich syndrome/X-linked thrombocytopenia: WASP gene mutations, protein expression, and phenotype. Blood. 1997 Oct 1;90(7):2680-9. PMID 9326235